CLINICAL TRIAL: NCT02777541
Title: Evaluation of Tolerance and Safety of Early Enteral Nutrition in Children After Percutaneous Endoscopic Gastrostomy Placement
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Children's Memorial Health Institute, Poland (Other)
Collaborators: Nutricia Foundation (Other)
Responsible Party: Principal Investigator, JAROSLAW KIERKUS, PhD, Children's Memorial Health Institute, Poland
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: RG 1/2014
Record Dates: First submitted 2016-05-16; First posted 2016-05-19 (Estimated); Last update posted 2016-05-20 (Estimated); Status verified 2016-05

CONDITIONS: Enteral Nutritional Support
Keywords: early enteral nutrition; children; percutaneous endoscopic gastrostomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Early enteral nutrition (Other): 3 hours after PEG implantation
  Interventions: Dietary Supplement: Resumption of feeding 3 hours after PEG placement
- Late enteral nutrition (Other): 8 hours after PEG implantation
  Interventions: Dietary Supplement: Resumption of feeding 8 hours after PEG placement

INTERVENTIONS:
Dietary Supplement: Resumption of feeding 3 hours after PEG placement — The first feeding will be with polymeric diet (1 kcal/ml). First feeding portion will have the volume equal to 1/3 of full recommended portion, volume of second feeding will be equal to 2/3 of full recommended portion and third portion will be equal to full recommended portion. Each portion will introduced thru the enteral feeding pump (Flocare Infinity, Nutricia), for 30 minutes, three-hour break between feeds. Infusion of 5% glucose solution with electrolytes will be given through intravenous line to cover maintenance fluid requirement in all subjects.
  Arms: Early enteral nutrition
Dietary Supplement: Resumption of feeding 8 hours after PEG placement — The first feeding will be with polymeric diet (1 kcal/ml). First feeding portion will have the volume equal to 1/3 of full recommended portion, volume of second feeding will be equal to 2/3 of full recommended portion and third portion will be equal to full recommended portion. Each portion will introduced thru the enteral feeding pump (Flocare Infinity, Nutricia), for 30 minutes, three-hour break between feeds. Infusion of 5% glucose solution with electrolytes will be given through intravenous line to cover maintenance fluid requirement in all subjects.
  Arms: Late enteral nutrition

SUMMARY:
There aren't sufficient randomized prospective controlled trials in pediatric population comparing the safety and tolerance of early feeding after PEG placement (3-4 hours). Most patients are fasted for at least 12 hours following percutaneous endoscopic gastrostomy. In order to decrease the period of fasting, inadequate nutritional support, and hospitalization time, the investigators decided to design this study. The additional goal is to establish an optimum standard procedure in the group of pediatric patients qualified for PEG insertion procedure in Poland.

DETAILED DESCRIPTION:
This study is a multicentre, randomized, open label trial designed to evaluate the tolerance and safety of early enteral nutrition after PEG placement in children. Recruitment will be from patients attending the one of six medical centers in Poland: Department of Gastroenterology, Hepatology and Feeding Disorders and Department of Pediatrics, The Children's Memorial Health Institute in Warsaw, Department of Pediatrics, Gastroenterology, Hepatology and Nutrition, Medical University of Gdańsk in Gdańsk, Department of Allergology, Gastroenterology and Nutrition, Medical University in Łódź, Department of Pediatrics, Medical University of Silesia in Katowice and Department of Pediatrics and Gastroenterology, Area Hospital in Torus.

The trial will include 100 patients, from 1-month-old to 18-year-old, qualified for percutaneous endoscopic gastrostomy (PEG) placement. All participants will be prepared for the procedure according to the standard medical protocol.

Parents/legal guardians, and where possible also the patient, will be informed about the research plan, and after signed informed consent to participate in the study patients will be enrolled for the study. At the Baseline visit participants will be randomized (1:1) to one of two treatment group: Group I- early enteral feeding group (3 hours after PEG implantation) or Group II- late enteral feeding group (8 hours after PEG implantation). The follow-up visits in hospital is planned 3, 6, 9 mad 12 months after the procedure in all subjects.

Primary endpoint:

1. Number of patients who will achieve full feed (total fluid and caloric requirements) within 48 hours since the first feeding bolus.

Secondary endpoints:

1. Number of early complications (to 6 days after PEG placement)
2. Number of late complications ( 7 days - 12 months after PEG placement)
3. Duration of hospitalization after PEG placement (in days)
4. Gastric residuals (ml) - sum up to 48 hours since the first feeding bolus

Tertiary endpoints:

1. Improvement in nutritional status (3,6,9,12 months after the procedure) - body weight gain (kg) and height gain (cm), BMI kg/m2
2. Influence of vitamin and trace element deficiency (vitamin D - 25(OH)D3, vitamin A, vitamin E, sodium, potassium, calcium, zinc, iron, magnesium, selenium) and other biochemical parameters abnormalities (serum level of urea, total protein, albumin, glucose, glycated hemoglobin (hemoglobin HbA1c), aspartate transaminase (AST), alanine transaminase (ALT), ferritin, C reactive protein) on complications rate.
3. Influence of ghrelin, leptin and adiponectin level on nutritional status improvement after PEG placement.
4. Influence of gastroesophageal reflux (GER) diagnosed before the procedure on feeding tolerance.
5. Corelation between fecal calprotectin level and feeding tolerance after PEG placement, complication rate and nutritional status before PEG placement.
6. Influence of oropharyngeal flora on complications rate (wound infection)
7. Correlation between PEG placement and GER.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects between 1 month-old and 18 years-old
2. Medical indications for percutaneous endoscopic gastrostomy (PEG) placement.
3. Informed consent to participate in the study signed and dated by the subject's parent/legal guardian and the also by patient over the age of 16 years.

Exclusion Criteria:

1. Serious, uncorrectable coagulation disorders.
2. Inability to perform upper gastrointestinal (UGI) series endoscopy (laryngeal or oesophageal stricture)
3. Need for concomitant fundoplication.
4. Lack of technical ability to perform PEG placement procedure

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-01; Primary Completion 2017-01 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients who will achieve full feed (total fluid and caloric requirements) within 48 hours since the first feeding bolus. | 48 hours

SECONDARY OUTCOMES:
Number of early complications (to 6 days after PEG placement) | to 6 days after PEG placement
Number of late complications ( 7 days - 12 months after PEG placement) | 7 days- 12 months after PEG placement
Number of hospitalization days after PEG placement | up to 30 days
Gastric residuals (ml) - sum up to 48 hours since the first feeding bolus | 48 hours

OTHER OUTCOMES:
Improvement in nutritional status | 12 months
  number of patients with nutritional status improvement after PEG placement
Influence of vitamin and trace element deficiency on complications rate. | 12 months
  number of patients with vitamin and trace deficiency before PEG placement who had diagnosed post PEG placement early or late complication.
Influence of ghrelin, leptin and adiponectin level on nutritional status | 12 months
  number of patients with incorrect ghrelin, leptin or adiponectin level with no post PEG nutritional improvement
Influence of gastroesophageal reflux (GER) diagnosed before the procedure on feeding tolerance. | 12 months
  number of patients with diagnosed pre PEG GER with no post PEG nutritional improvement
Corelation between fecal calprotectin level and feeding tolerance after PEG placement | 12 months
  number of patients with elevated calprotectin level before PEG placement who had post PEG placement enteral feeding intolerance
Influence of oropharyngeal flora on complications rate (wound infection) | 12 months
  number of patients with abnormal oropharyngeal flora with post PEG wound infection
Correlation between PEG placement and GER | 12 months
  number of patients with post PEG GER

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Gastroenterology, Hepatology and Feeding Disorders, Warsaw, Poland

REFERENCES:
- [Derived] Wiernicka A, Matuszczyk M, Szlagatys-Sidorkiewicz A, Landowski P, Toporowska-Kowalska E, Gebora-Kowalska B, Popinska K, Sibilska M, Grzybowska-Chlebowczyk U, Wiecek S, Hapyn E, Blimke-Koziel K, Kierkus J. Tolerability and safety of early enteral nutrition in children after percutaneous endoscopic gastrostomy placement: A multicentre randomised controlled trial. Clin Nutr. 2019 Aug;38(4):1544-1548. doi: 10.1016/j.clnu.2018.08.018. Epub 2018 Aug 28. PMID 30197271
- [Derived] Wiernicka A, Matuszczyk M, Szlagatys-Sidorkiewicz A, Toporowska-Kowalska E, Popinska K, Chlebowczyk-Grzybowska U, Hapyn E, Kierkus J. The protocol for a randomised-controlled trial of the evaluation of the tolerance and safety of early enteral nutrition in children after percutaneous endoscopic gastrostomy placement. (protocol version 09.01.2015). BMC Pediatr. 2016 Oct 7;16(1):163. doi: 10.1186/s12887-016-0705-8. PMID 27717336